CLINICAL TRIAL: NCT07369726
Title: The Effect of Early Post-Cesarean Mobilization and Caffeine Consumption on Bowel Motility, Pain, and Psychological Well-being: A Randomized Controlled Trial
Brief Title: Effects of Mobilization and Caffeine After Cesarean
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Hafize Dağ Tüzmen, DOCTORAL PROFESSOR, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AIBU-EBE-EK-01
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Gastrointestinal Motility; Postoperative Pain; Psychological Well-Being
Keywords: gastrointestinal motility; postoperatif pain; Psychological Well-Being; Early Ambulation
MeSH Terms: conditions — Pain, Postoperative; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Women in the control group will receive routine intervention. They will be mobilized at 6 hours. Decaffeinated coffee will be served at 6-hour intervals.
  Interventions: Dietary Supplement: Decaffeinated coffee
- intervention group (Experimental): They will be mobilized at 4 hours.They will consume Turkish coffee containing caffeine every six hours.
  Interventions: Dietary Supplement: caffeine consumption

INTERVENTIONS:
Dietary Supplement: caffeine consumption — The women in the intervention group will be mobilised at the 4-hour mark. The intervention group will be given caffeinated Turkish coffee at 6-hour intervals.
  Arms: intervention group
Dietary Supplement: Decaffeinated coffee — The women in the control group will be mobilised at the 6-hour mark. The control group will be given decaffeinated Turkish coffee at 6-hour intervals.
  Arms: Control Group

SUMMARY:
This study Maims to assess bowel motility, pain and psychological well-being in women in the post-cesarean period by mobilizing them early and encouraging them to consume coffee.

DETAILED DESCRIPTION:
In the intervention group, the goal is to initiate bowel motility by mobilizing women early in the post-cesarean period. This increased bowel motility will facilitate gas expulsion, thus minimizing pain levels. Caffeine consumption will help keep pain levels at a minimum. By minimizing pain, women will experience positive psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Being between 18 and 35 years of age,
2. Women who underwent cesarean delivery under spinal anesthesia,
3. Having a post-cesarean pain level of 4 or higher,
4. Being able to understand and write Turkish and communicate effectively with researchers.

Exclusion Criteria:

1. Women who underwent emergency cesarean delivery,
2. Those with pregnancy complications (preeclampsia, placenta previa, etc.),
3. Those with a history of chronic gastrointestinal disease (e.g., irritable bowel syndrome, Crohn's disease, ulcerative colitis),
4. Those with sensitivity or allergy to caffeine,
5. Those with a history of chronic pain syndrome or dependence on analgesics,
6. Regular coffee drinkers (≥2 cups per day),
7. Intraoperative complications such as bowel or bladder injury,

i) Those who cannot comply with the study protocol or complete the follow-up process.

Removal Criteria:

1. Participants are excluded from the study under the following conditions:
2. During surgery If complications occur (e.g., bladder or bowel injury, excessive bleeding),
3. Postoperative complications requiring admission to the intensive care unit (ICU) for the mother or newborn,
4. Development of severe postoperative nausea, vomiting, or intolerance to oral intake,
5. Inability to consume or refusal to consume coffee according to the study protocol,
6. Withdrawal of consent by the participant at any point during the study,
7. Failure to comply with surgical procedures or loss of follow-up,
8. Development of medical conditions during follow-up that may affect study results (e.g., acute infections, neurological disorders).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women aged 18-35
Enrollment: 60 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in postoperative pain after caesarean section within 24 hours from baseline | Starting point, after intervention at 6 hours, 12 hours, 18 hours and 24 hours
  Pain will be assessed using a 10 cm visual analogue scale. '0' means no pain, while '10' means unbearable pain. The assessment will be carried out at the start of the study, at 6-hour intervals, and at the end.
Change in postoperative Bowel Motility after caesarean section within 24 hours from baseline | Starting point, after intervention at 6 hours, 12 hours, 18 hours and 24 hours
  Bowel motility will be assessed using BFI. The Bowel Function Index (BFI) is a short and practical measure used to assess constipation, particularly in patients using opioids. It consists of three questions, each scored on a scale of 0 to 100. These scores are used to measure the degree of bowel dysfunction.
Change in postoperative Psychological Well-being after caesarean section within 24 hours from baseline | Starting point, after intervention at 6 hours, 12 hours, 18 hours and 24 hours
  Psychological Well-being will be assessed using Psychological Well-Being Scale. Based on the score obtained: 1.00-2.99 → Low psychological resilience, 3.00-4.30 → Moderate level, 4.31-5.00 → High psychological resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No